CLINICAL TRIAL: NCT01080183
Title: Functional Assessment Screening Tablets - Patient Reported Measures Translating Research Into Practice Pilot
Brief Title: Functional Assessment Screening Tablets - Patient Reported Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: RAND (Other)
Responsible Party: Principal Investigator, Rachel Hess, MD, MS, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO09080140
Record Dates: First submitted 2010-02-27; First posted 2010-03-03 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Smoking
Keywords: Health-related quality of life; physical activity
MeSH Terms: conditions — Smoking; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback form (Experimental): patients receive feedback regarding their prms in addition to doctor receiving report
  Interventions: Other: Patient feedback form
- usual care (No Intervention): patients do not receive feedback form prior to the encounter, clinicians continue to receive patient reported measures prior to the appointment

INTERVENTIONS:
Other: Patient feedback form — patients receive a report that feeds back their patient reported measures to them prior to their clinical visit
  Arms: Feedback form

SUMMARY:
The team's ultimate goal is to improve health care quality and effectiveness and support patient-centered care. In this project, we, the investigators, will test whether providing patients with guideline based-recommendations regarding tobacco use, physical activity and mental and physical health-related quality of life (patient reported measures: PRMs) using health information technology increases doctor-patient discussions regarding these topics and results in improvements in PRMs. We will randomize physicians in a single general internal medicine practice. Patients seeing intervention physicians will receive guideline-based recommendations regarding PRMs, those seeing control physicians will not. We will compare differences in doctor-patient discussions regarding PRMs between the intervention and control groups. The successful completion of this project will provide evidence the effectiveness of involving patients in their care through the use guideline-based feedback.

ELIGIBILITY:
Inclusion Criteria:

* physicians who see patients in the University of Pittsburgh General Internal Medicine Practice.
* patients of physician's who have consented to participate.

Exclusion Criteria:

* age less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Doctor Patient Communication | The doctor and patient pair will complete a one time survey within two weeks of the doctor patient encounter. Audiotaping of the encounter will occur once at the time of encounter.
  the doctor patient and encounter will be queried for communication regarding the patient reported measures

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hess, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- General Internal Medicine Oakland, Pittsburgh, Pennsylvania, United States